CLINICAL TRIAL: NCT05701501
Title: Clinical Study of Vitamin B5 in Adjuvant Treatment of Inflammatory Bowel Disease
Brief Title: Clinical Study of Vitamin B5 in Adjuvant Treatment of IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: The University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of gastroenterology department, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VitB5
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Vitamin B5,treatment
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Pantothenic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B5 group (Experimental): Based on the standard IBD treatment, Vitamin B5 (5mg/tablet) is given orally three times a day, four tablets each time, for 12 weeks.
  Interventions: Drug: Vitamin B5 Tablets
- Control group (Placebo Comparator): Based on the standard IBD treatment, the same type of placebo tablets are given orally three times a day, four tablets each time, for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin B5 Tablets — The experimental group was given Vitamin tablets (5mg/tablet) based on the standard IBD treatment.
  Arms: Vitamin B5 group
Drug: placebo — The control group was given placebo tablets of the same type based on the standard IBD treatment.
  Arms: Control group

SUMMARY:
Patients with IBD are randomized to oral administration of vitamin B5 and placebo based on the standard treatment, exploring whether Vitamin B5 can increase the clinical remission rate of IBD patients and improve the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBD according to the consensus on the diagnosis and treatment of inflammatory bowel disease (Beijing, 2018, DOI:10.19538/j.nk2018090106);
* Have complete medical history data;
* Volunteer to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* Hemophilic patients;
* There are abdominal abscesses, toxic megacolon, fulminant colitis, partial colectomy, or total colectomy;
* Other autoimmune diseases, hematological diseases, tumors, acute infection, severe liver and kidney insufficiency, serious diseases such as severe anemia, neutropenia, heart failure, organic heart disease, hepatitis B, liver cirrhosis, kidney disease and mental diseases;
* Take calcium pantothenate preparation in recent 3 months;
* Have a history of abuse of psychoactive substances;
* Pregnant or lactating women, or plan to be pregnant in the next 6 months;
* Nervous system diseases: such as Alzheimer's disease, stroke, Parkinson's disease;
* Participate in other clinical trials in the past 6 months;
* Incomplete medical record information (including gender, age, diagnosis information, colonoscopy results, pathological diagnosis results and other demographic data)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | Through study completion, an average of 12 months.
  To evaluate the improvement effect of clinical remission rate (Mayo score ≤ 2 points and no single sub-score>1 point; CDAI score<150) in IBD patients after 12 weeks of oral Vitamin B5 while taking routine treatment.

SECONDARY OUTCOMES:
Disease activity score of IBD patients | Through study completion, an average of 12 months.
  Modified Mayo score or CDAI score
Histological remission | Through study completion, an average of 12 months.
  Based on the Geboes scale. No or slight increase of chronic inflammatory infiltration in lamina propria, no neutrophils in lamina propria or epithelium, no persistent clinical response of erosion, ulcer or granulation tissue.
Clinical response | Through study completion, an average of 12 months.
  Modified Mayo score decreased by 2 points and 30% from baseline+rectal bleeding score decreased by 1 point or absolute rectal bleeding score decreased by 1 point.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital; Shu Zhu, PhD, Study Director — The University of Science and Technology of China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No